CLINICAL TRIAL: NCT00331006
Title: Rituximab for the Treatment of Inhibitors in Congenital Hemophilia A (A TMH CTN Study)
Brief Title: Rituximab to Treat Severe Hemophilia A
Acronym: RICH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Carelon Research (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 374; U01HL072268 (NIH); U01HL072274 (NIH); U01HL072290 (NIH); U01HL072033 (NIH); U01HL072291 (NIH); U01HL072248 (NIH); U01HL072355 (NIH); U01HL072283 (NIH); U01HL072346 (NIH); U01HL072331 (NIH)
Record Dates: First submitted 2006-05-26; First posted 2006-05-29 (Estimated); Results first posted 2013-06-11 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Hemophilia A
Keywords: Blood Coagulation Factor Inhibitors
MeSH Terms: conditions — Hemophilia A | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rituximab (Experimental): Rituximab administered at a dose of 375 mg/m2 by slow intravenous infusion once per week for 4 weeks
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Rituximab by slow intravenous infusion; for participants greater than or equal to 10 kg, 375 mg per m^2 BSA weekly for 4 weeks; for participants less than 10 kg, 12.5 mg/kg weekly for 4 weeks
  Other Names: Rituxan

SUMMARY:
Hemophilia A is a serious blood clotting disorder caused by a lack of factor VIII, a specialized protein needed for normal blood clotting to occur. Individuals with this disease may experience spontaneous bleeding, pain and swelling in their joints due to excess bleeding, and bruising. A common treatment for severe hemophilia A is to intravenously replace the deficient blood clotting factor; however, some individuals may develop antibodies to this replacement factor. This study will evaluate the effectiveness of rituximab at reducing the antibodies that develop in response to the replacement factor in individuals with severe hemophilia A.

DETAILED DESCRIPTION:
Hemophilia A is a hereditary blood clotting disorder. It is caused by a deficiency or abnormality of the blood clotting protein factor VIII. Individuals with hemophilia A are unable to form blood clots to stop bleeding and are at risk for experiencing serious and life-threatening bleeding episodes. The most common treatment for this disease is intravenous replacement of factor VIII. However, between 30 to 40% of individuals eventually develop inhibitors, or antibodies, to the replacement factor. In these individuals, the immune system recognizes the replacement factor as foreign and attacks it, thereby countering any potential benefits of the treatment. Some individuals with severe hemophilia A may undergo immune tolerance therapy (ITT), in which they receive replacement factor on a regular basis as a way for the body to adjust to the factor and stop inhibitor production. This treatment, however, is not always effective for everyone. Preliminary research has shown that rituximab, a medication used to treat non-Hodgkin's lymphoma, may be successful in suppressing or eliminating the inhibitors that develop. The purpose of this study is to evaluate the effectiveness of rituximab at lowering the levels of factor VIII inhibitors in individuals with severe hemophilia A.

This study will enroll individuals with severe hemophilia A. At study entry, participants will receive one intravenous dose of factor VIII. Inhibitor levels will be measured with a blood test 5 to 7 days following this procedure. If peak inhibitor level is above 5 Bethesda units (BU)/mL, 5 to 9 days later participants will begin receiving rituximab intravenously once a week for 4 weeks. Blood will be collected at each visit for laboratory testing. Two weeks following the last rituximab treatment, participants will have blood drawn for inhibitor testing; this testing will occur every 4 weeks through Week 22. If the participant's inhibitor level falls below 5 BU/mL, participants will receive a repeat dose of factor VIII, and blood will be drawn 5 to 7 days later for inhibitor testing. Follow-up visits will occur at Weeks 36, 52, and 100, and will include a physical examination, blood collection, and monitoring of bleeding events and infections. Telephone interviews will be conduced at Weeks 64, 76, and 88 to monitor bleeding events and infections.

ELIGIBILITY:
Inclusion Criteria:

* Severe congenital hemophilia A
* Documented historical inhibitor titer to factor VIII of at least 5 BU/mL
* Inhibitor level greater than or equal to 5 BU/mL 5 to 14 days after initial factor VIII exposure during screening

Exclusion Criteria:

* Known hypersensitivities or allergies to murine and/or humanized antibodies
* Currently participating in investigational hemophilia studies
* HIV infected
* Any immunodeficiency disorder
* Liver disease and serum ALT or AST is greater than three times the upper limit of normal, albumin is less than 2.5g/dl, and/or INR is greater than 1.7
* Received interferon or other immunomodulatory drugs, such as steroids or cytotoxic therapy in the 30 days prior to study entry
* History of cardiac arrhythmias, any active febrile illness, kidney insufficiency, or pulmonary infiltrates
* Has previously received rituximab treatment
* Currently undergoing immune tolerance therapy
* Evidence of Hepatitis B (HBV) infection, defined as one of the following:

  * HBsAg positive
  * HBsAg negative, HBsAb negative, HBcAb positive, and HBV DNA positive
* Participants with a high responding inhibitor (at least 5 BU/mL) first detected fewer than 12 months prior to study entry, unless the participant has failed immune tolerance therapy, defined as one of the following:

  1. Failure to fulfill the criteria for full or partial success within 33 months, as defined by a factor VIII recovery greater than or equal to 66% of expected and half-life greater than or equal to 6 hours measured after a 72-hour treatment-free washout period
  2. Failure to achieve greater than 20% reduction in inhibitor titer during each interim non-overlapping 6-month period of ITT in the absence of documented infection, with 9 months as the minimum treatment period and 33 months as the maximum possible duration of unsuccessful ITT
  3. Withdrawal from ITT for any other reason
* Routinely receive factor VIII concentrate for the treatment of both major and minor bleeding events
* Has received factor VIII concentrate in the 7 days prior to study entry

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2006-06; Primary Completion 2010-11 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan F. Assmann, PhD, Principal Investigator — NERI; Cindy Leissinger, MD, Principal Investigator — Tulane University Health Sciences Center; Joan Gill, MD, Principal Investigator — Versiti Blood Health; Keith McCrae, MD, Principal Investigator — University Hospital of Cleveland; Ellis Neufeld, MD, Principal Investigator — Boston Children's Hospital; Cassandra Josephson, MD, Principal Investigator — Children's Healthcare of Atlanta; Nigel Key, MD, Principal Investigator — University of North Carolina; Charles Sexauer, MD, Principal Investigator — University of Oklahoma; Janna Journeycake, MD, Principal Investigator — University of Texas Southwestern Medical Center; Leslie Raffini, MD, Principal Investigator — Children's Hospital of Philadelphia; Margaret Ragni, MD, Principal Investigator — Hemophilia Center of Western Pennsylvania; Leonard Valentino, MD, Principal Investigator — Rush University Medical Center; Diane Nugent, MD, Principal Investigator — Children's Hospital of Orange County; Marcella Torres, MD, Principal Investigator — Cook Children's Medical Center
Locations (13):
- United States (13):
  - Children's Hospital of Orange County, Orange, California
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Children's Hospital Boston, Boston, Massachusetts
  - UNC at Chapel Hill Hospital, Chapel Hill, North Carolina
  - University Hospital of Cleveland, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Hemophilia Center of Western Pennsylvania, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Comprehensive Center for Bleeding Disorders, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at clinical sites and Hemophilia Treatment Centers participating in the study. The recruitment period began in August 2006 and continued through November 2011.
Groups:
- Rituximab: Rituximab administered at a dose of 375 mg/m^2 by slow intravenous infusion once per week for 4 weeks
Period: Screening Phase
Arm/Group | Rituximab
Started | 23
Completed | 16 (subjects eligible for the treatment phase if inhibitor titer following Factor VIII was at least 5 BU)
Not Completed | 7
Not completed — Withdrawal by Subject | 1
Not completed — enrollment halted | 1
Not completed — Lost to Follow-up | 1
Not completed — Ineligible for treatment phase | 4
Period: Treatment Phase
Arm/Group | Rituximab
Started | 16
Completed | 15
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Follow-Up Phase I
Arm/Group | Rituximab
Started | 15
Completed | 14
Not Completed | 1
Not completed — Lost to Follow-up | 1
Period: Follow-Up Phase II
Arm/Group | Rituximab
Started | 14
Completed | 11
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Population: All subjects who began the screening phase
Arm/Group | Rituximab
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 19
  Between 18 and 65 years | 4
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 15.85 (12.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 23
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With Major Response, i.e. Inhibitor Level Falls to Less Than 5 BU/mL Between Weeks 6 to 22 and Remains Below 5 BU/mL at 5-7 Days Following Re-challenge With FVIII
Description: Presence or absence of a major response in each participant. Major response is defined as occurring when inhibitor level falls to less than 5 BU/mL between Weeks 6 to 22 and remains below 5 BU/mL at 5-7 days following re-challenge with FVIII
Time Frame: Measured within approximately 22 weeks
Population: All participants who received at least one dose of rituximab
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Rituximab
Number analyzed (Participants) | 16
proportion of participants | .1875 [0.053 to 1.0]
Statistical Analysis 1: Comparison: Rituximab; The null hypothesis is that the proportion of participants in which the inhibitor level falls to less than 5 BU/mL between weeks 6 to 22 and remains below 5 BU/mL at 5-7 days following re-challenge with factor VIII is no more than 0.05; Test type: Superiority or Other; p = 0.043, Exact Binomial — the a priori p-value was 0.05 for statistical significance; Proportion = .1875, 95% CI 1-sided [lower limit .053]

2. Secondary Outcome: Proportion of Subjects With at Least Minor Response, i.e. Inhibitor Level Falls to <5 BU/mL Between Weeks 6-22 and Either Remains <5 BU/mL 5-7 Days Following FVIII Rechallenge or Titer Following FVIII Rechallenge is 5-10 BU/mL & <50% of Original Peak
Description: Presence or absence of at least a minor response in each participant
Time Frame: Measured within approximately 22 weeks
Population: All participants who received at least one dose of rituximab
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Rituximab
Number analyzed (Participants) | 16
proportion of participants | 0.25 [0.073 to 0.524]
Statistical Analysis 1: Comparison: Rituximab; No hypothesis about the value of this proportion was specified in the study design; Test type: Superiority or Other; Exact Binomial; Proportion = .25, 95% CI 2-sided [0.073 to 0.524]

3. Secondary Outcome: Percent Change in Inhibitor Titer on Challenge With Factor VIII From Baseline Challenge to Post-treatment Challenge
Description: percent change=100%*(A-B)/B where A=inhibitor titer measured within 5-7 days following FVIII rechallenge and B=inhibitor titer measured within 5-14 days following baseline FVIII challenge. A FVIII rechallenge was performed within 10-18 days of the first monthly study visit in which an inhibitor titer result <5 BU/mL was obtained beginning 2 weeks and continuing through 18 weeks following the last rituximab infusion.
Time Frame: Measured within approximately 22 weeks
Population: All subjects who received a post-treatment rechallenge and had at least a minor response.
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | Rituximab
Number analyzed (Participants) | 4
percentage change | -64.31 [-77.11 to -44.49]

4. Secondary Outcome: Median Number of Bleeding Events Per Subject Meeting the Criteria of a Serious Adverse Event
Description: Median number of bleeding events per subject meeting the criteria of a serious adverse event
Time Frame: Measured through Week 100
Population: Data on bleeding events were collected at every study visit for all study participants. Data for this outcome was collected through the particpants end of study or Week 100, whichever came first, and is restricted to the 16 subjects who received at least one dose of rituximab.
Measure: Median (Inter-Quartile Range); unit: participants
Arm/Group | Rituximab
Number analyzed (Participants) | 16
participants | 0 [0 to 2]

5. Secondary Outcome: Median Number of Bleeding Events Per Subject Not Meeting the Criteria of a Serious Adverse Event
Description: Median Number of Bleeding Events Per Subject Not Meeting the Criteria of a Serious Adverse Event
Time Frame: Measured through Week 100
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: participants
Arm/Group | Rituximab
Number analyzed (Participants) | 16
participants | 19.5 [11 to 41]

6. Secondary Outcome: Median Number of Serious Adverse Events Per Subject Other Than Bleeding Events
Description: Median Number of Serious Adverse Events Per Subject Other Than Bleeding Events
Time Frame: Measured through Week 100
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: participants
Arm/Group | Rituximab
Number analyzed (Participants) | 16
participants | 1 [0 to 2.5]

7. Secondary Outcome: Median Number of Adverse Events Per Subject That Were Not Bleeding Events and Did Not Meet the Criteria of a Serious Adverse Event
Description: Median Number of Adverse Events Per Subject That Were Not Bleeding Events and Did Not Meet the Criteria of a Serious Adverse Event
Time Frame: Measured through Week 100
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: participants
Arm/Group | Rituximab
Number analyzed (Participants) | 16
participants | 1.5 [0 to 4]

8. Secondary Outcome: Proportion of Rituximab Infusions in Which a Reaction to the Infusion Was Reported
Description: Proportion of rituximab infusions in which a reaction to the infusion was reported
Time Frame: Measured at Week 1 through Week 4
Population: All rituximab infusions given to study participants
Measure: Number (95% Confidence Interval); unit: proportion of rituximab infusions
Units Other Than Participants: rituximab infusions
Arm/Group | Rituximab
Number analyzed (Participants) | 16
Number analyzed (rituximab infusions) | 61
proportion of rituximab infusions | 0.11 [0.05 to 0.22]

ADVERSE EVENTS:
Time Frame: Through week 100
Description: Restricted to the 16 subjects who received at least one dose of rituximab.
Arm/Group | Rituximab
Serious Adverse Events (participants affected / at risk) | 11/16
Other Adverse Events (participants affected / at risk) | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab (N=16)
Diarrhea (Gastrointestinal disorders) | 1 (1) — Meeting Serious Adverse Event Criteria
Mallory-Weiss tear (Gastrointestinal disorders) | 1 (1)
Allergic reaction/hypersensitivity (General disorders) | 1 (1)
Fever (General disorders) | 1 (1) — Meeting Serious Adverse Event Criteria
Central line infection (Infections and infestations) | 1 (1)
Pulmonary/upper respiratory infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Viral meningitis (Infections and infestations) | 1 (1)
Zoster infection (Infections and infestations) | 1 (1)
Bleeding and/or hematoma due to injury (Injury, poisoning and procedural complications) | 1 (1) — Meeting serious adverse event criteria
Bleeding and/or hematoma due to procedure complication (Injury, poisoning and procedural complications) | 1 (1) — Meeting serious adverse event criteria
Hematoma due to injury (Injury, poisoning and procedural complications) | 1 (2) — Meeting serious adverse event criteria
Hematoma due to procedure complication (Injury, poisoning and procedural complications) | 1 (1) — Meeting serious adverse event criteria
Joint and other bleeding due to injury (Injury, poisoning and procedural complications) | 1 (2) — Meeting serious adverse event criteria
Joint bleeding due to injury (Injury, poisoning and procedural complications) | 3 (6) — Meeting serious adverse event criteria
Bleeding and/or hematoma - spontaneous (Musculoskeletal and connective tissue disorders) | 1 (1) — Meeting serious adverse event criteria
Bone fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint and other bleeding - spontaneous (Musculoskeletal and connective tissue disorders) | 1 (1) — Meeting serious adverse event criteria
Joint bleeding - spontaneous (Musculoskeletal and connective tissue disorders) | 4 (11) — Meeting serious adverse event criteria
Joint bleeding due to procedure complication (Injury, poisoning and procedural complications) | 1 (1)
Headache (Nervous system disorders) | 1 (1) — Meeting serious adverse event criteria
Subdural hemorrhage (Nervous system disorders) | 1 (2)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Meeting serious adverse event criteria
Port placement (Surgical and medical procedures) | 1 (1)
Port removal and replacement (Surgical and medical procedures) | 1 (1)
Synovectomy (Surgical and medical procedures) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) — Meeting serious adverse event criteria
Splenic hematoma (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab (N=16)
Anemia (Blood and lymphatic system disorders) | 1 (3)
Enlarged lymph nodes (Blood and lymphatic system disorders) | 1 (1)
Increased blood lymphocytes (Blood and lymphatic system disorders) | 1 (1)
Increased blood monocytes (Blood and lymphatic system disorders) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
White blood cell decrease (Blood and lymphatic system disorders) | 1 (3)
Sweating (Endocrine disorders) | 1 (1)
Pink eye (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (3)
Bleeding - spontaneous (Gastrointestinal disorders) | 4 (12)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Heartburn (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (3)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (4)
Bleed and/or hematoma (General disorders) | 1 (1)
Chills (General disorders) | 3 (3)
fatigue (General disorders) | 1 (2)
Fever (General disorders) | 2 (4)
Lethargy (General disorders) | 1 (1)
Decreased ALT (Hepatobiliary disorders) | 1 (3)
Elevated ALT (Hepatobiliary disorders) | 1 (7)
Allergy (Immune system disorders) | 1 (1)
Cold sore (Infections and infestations) | 1 (1)
Group A strep (Infections and infestations) | 1 (2)
Influenza (Infections and infestations) | 2 (2)
Septic polyarthritis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Bleed and/or hematoma due to injury (Injury, poisoning and procedural complications) | 4 (12)
Bleeding due to injury (Injury, poisoning and procedural complications) | 3 (9)
Bleeding due to procedure complication (Injury, poisoning and procedural complications) | 2 (2)
Head injury (Injury, poisoning and procedural complications) | 2 (2)
Joint bleeding due to injury (Injury, poisoning and procedural complications) | 11 (31)
Joint pain due to injury (Injury, poisoning and procedural complications) | 1 (1)
vaccination site reaction (Injury, poisoning and procedural complications) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Joint bleeding, spontaneous (Musculoskeletal and connective tissue disorders) | 15 (262)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint pain, spontaneous (Musculoskeletal and connective tissue disorders) | 1 (2)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle pain, spontaneous (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bleed and/or hematoma - spontaneous (Musculoskeletal and connective tissue disorders) | 10 (26)
Bells palsy (Nervous system disorders) | 1 (1)
Bleeding - spontaneous (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Intolerance to light (Nervous system disorders) | 1 (1)
Bleeding - spontaneous (Renal and urinary disorders) | 1 (2)
Hematuria (Renal and urinary disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Bleeding - spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cold (Reproductive system and breast disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Elevated carbon dioxide in the blood (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Runny nose (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Bleed and/or hematoma - spontaneous (Skin and subcutaneous tissue disorders) | 7 (20)
Hematoma - spontaneous (Skin and subcutaneous tissue disorders) | 9 (24)
Rash (Skin and subcutaneous tissue disorders) | 2 (3)
Sunburn (Skin and subcutaneous tissue disorders) | 1 (1)
High blood pressure (Vascular disorders) | 1 (1)
Low blood pressure (Vascular disorders) | 1 (4)
Pulmonary hypertension (Vascular disorders) | 1 (1)
Hematoma due to injury (Injury, poisoning and procedural complications) | 6 (14)
Hematoma due to procedure complication (Injury, poisoning and procedural complications) | 4 (5)
Pain (Injury, poisoning and procedural complications) | 1 (1)
Bleeding - spontaneous (Musculoskeletal and connective tissue disorders) | 1 (1)
Hematoma - spontaneous (Musculoskeletal and connective tissue disorders) | 3 (3)
Bleeding - spontaneous (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated before reaching its target sample size of 50 subjects due to low enrollment rates. Therefore, confidence intervals for proportions are wide.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Baxter donated Factor VIII and Genentech donated rituximab for the study. Both Baxter and Genentech can review results communications prior to public release for a period of time less than or equal to 60 days from the time submitted to them for review. These companies cannot require changes to the communication.